CLINICAL TRIAL: NCT03255187
Title: Effect of Dietary Supplementation With Fish Oil in Alleviating Cardiopulmonary Hazards Associated With Air Pollution
Brief Title: Effect of Dietary Supplemental Fish Oil in Alleviating Health Hazards Associated With Air Pollution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haidong Kan, PhD and Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FDUEH-3
Record Dates: First submitted 2017-08-12; First posted 2017-08-21 (Actual); Results first posted 2020-01-21 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Oxidative Stress; Inflammation; Blood Pressure; Vasoconstriction; Coagulation; Pulmonary Function
Keywords: Biomarker; Fish oil; Oxidative stress; Air pollution; Cardiopulmonary system
MeSH Terms: conditions — Inflammation; Thrombosis

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to two parallel groups at enrollment using a random-number table. And the investigators randomly assign the two groups in a double-blind fashion receive either ﬁsh oil or sunflower seed oil for 4 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fish oil supplementation (Experimental): This group receive 2.5 g/day (two 1.25-g capsules daily) of fish oil (marine-derived n-3 PUFA) for 4 consecutive months.
  Interventions: Dietary Supplement: Fish oil supplementation
- Sunflower seed oil supplementation (Placebo Comparator): This group receive 2.5 g/day (two 1.25-g capsules daily) of placebo (sunflower seed oil) for 4 consecutive months.
  Interventions: Dietary Supplement: Sunflower seed oil supplementation

INTERVENTIONS:
Dietary Supplement: Fish oil supplementation — Participants of this randomized double-blind placebo-controlled trial include 70 healthy Chinese adults. The investigators randomly assign participants to two parallel groups at baseline using a random-number table. Compliance is determined by directly observed supplement intake. Participants in fish oil group are assigned to receive 2.5 g/day in divided doses. Each capsule contains 60% n-3 PUFA [24% docosahexanoic acid (C22:6 n-3 DHA) and 36% eicosapentaenoic acid (C20:5 n-3 EPA)].
  Arms: Fish oil supplementation
Dietary Supplement: Sunflower seed oil supplementation — Participants of this randomized double-blind placebo-controlled trial include 70 healthy Chinese adults. The investigators randomly assign participants to two parallel groups at baseline using a random-number table. Compliance is determined by directly observed supplement intake. Participants in sunflower seed oil group receive 2.5 g/day in divided doses, and the capsules are identical as the fish oil capsules.
  Arms: Sunflower seed oil supplementation

SUMMARY:
This study aims to evaluate whether dietary supplementation with fish oil can protect against the cardiopulmonary alterations linked to air pollution

DETAILED DESCRIPTION:
The investigators conduct a randomized controlled trial among 70 healthy college students in Shanghai, China. These students fulfilling the recruitment criteria will be randomly divided into two parallel groups to receive either fish oil [marine-derived n-3 polyunsaturated fatty acids (PUFA)] or sunflower seed oil. Participants in fish oil group receive 2.5 g/day (two 1.25-g capsules daily) in divided doses. The sunflower seed oil capsules are identical. All interventions started at 7:30 a.m.to avoid issues related to diurnal variation. Health endpoints, including blood pressure, skin color, fractional exhaled nitric oxide and pulmonary function were evaluated and biological samples such as morning urine, fast blood, saliva sample,buccal cells and skin tape stripping will be collected at week 1 before supplemenatation, and week 8, week 10, week 12 as well as week 14 during the supplementation phase.The investigators measure personal real-time exposure to PM2.5 and personal temperature and relative humidity.

ELIGIBILITY:
Inclusion Criteria:

* Equal to or older than 18 years old.
* No history of smoking and alcohol addiction.
* No chronic diseases or respiratory or allergic diseases,such as hypertension,diabetes,chronic obstructive pulmonary disease,other respiratory/cardiovascular diseases, asthma, rhinitis or other allergic diseases reported by volunteers.
* No allergies to n-3 PUFA or fish.

Exclusion Criteria:

* Current smokers or ever smokers
* Chronic drug use due on cardiovascular or respiratory diseases
* Participants are taking fish oil,anti-inflammatory drugs, or antioxidant supplements (such as vitamin C or vitamin E)

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-09-09 (Actual); Primary Completion 2018-01-13 (Actual); Study Completion 2018-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haidong Kan, Study Director — School of Public Health，Fudan University
Locations (1):
- Department of Environmental Health, School of Public Health, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhou L, Jiang Y, Lin Z, Chen R, Niu Y, Kan H. Mechanistic insights into the health benefits of fish-oil supplementation against fine particulate matter air pollution: a randomized controlled trial. Environ Health. 2022 Oct 29;21(1):104. doi: 10.1186/s12940-022-00908-1. PMID 36309727
- [Derived] Lin Z, Chen R, Jiang Y, Xia Y, Niu Y, Wang C, Liu C, Chen C, Ge Y, Wang W, Yin G, Cai J, Clement V, Xu X, Chen B, Chen H, Kan H. Cardiovascular Benefits of Fish-Oil Supplementation Against Fine Particulate Air Pollution in China. J Am Coll Cardiol. 2019 Apr 30;73(16):2076-2085. doi: 10.1016/j.jacc.2018.12.093. PMID 31023432

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted on Agust, 2017 in Fenglin Campus, Fudan University. A total of 93 participants were assessed for eligibility and 70 of them were finally recruited.
Groups:
- Sunflower Seed Oil Supplementation: This group receive 2.5 g/day (two 1.25-g capsules daily) of placebo (sunflower seed oil) for 4 consecutive months.
  Sunflower seed oil supplementation: Participants of this randomized double-blind placebo-controlled trial include 70 healthy Chinese adults. The investigators randomly assign participants to two parallel groups at baseline using a random-number table. Compliance is determined by directly observed supplement intake. Participants in sunflower seed oil group receive 2.5 g/day in divided doses, and the capsules are identical as the fish oil capsules. Each capsule containes 14.4% palmitic acid (C16:0), 16.0% oleic acid (C18:1 n-9), and 57.6% linoleic acid (C18:2 n-6).
Period: Periodfrom Enrollment to First Follow-up
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
Started | 35 | 35
Completed | 34 | 32
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3
Period: Period From First to Second Follow-up
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
Started | 34 | 32
Completed | 34 | 31
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Period From Second to Third Follow-up
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
Started | 34 | 31
Completed | 34 | 31
Not Completed | 0 | 0
Period: Period From Third to Fourth Follow-up
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
Started | 34 | 31
Completed | 34 | 31
Not Completed | 0 | 0
Period: Period at Fourth Follow-up
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
Started | 34 | 31
Completed | 34 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation | Total
Number analyzed (Participants) | 34 | 31 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.03 (2.26) | 22.87 (1.28) | 22.95 (1.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 14 | 13 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 34 | 31 | 65
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 34 | 31 | 65
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 21.73 (3.23) | 21.56 (3.02) | 21.65 (3.10)
Physical activity [Count of Participants; unit: Participants] — Physical activity: mild, 90-180 minutes/week; moderate, 180-360 minutes/week; and vigorous, >360 minutes/week.
  Participants
    Never | 31 | 27 | 58
    Mild | 2 | 3 | 5
    Moderate | 1 | 1 | 2
    Vigorous | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Biomarkers of Antioxidant Activity-Total Antioxidant Capacity (TAC) and Superoxide Dismutase (SOD)
Description: Peripheral blood samples (5 ml) were drawn, separated into serum, and stored at -80 ℃ within 30 minutes. We measure 2 biomarkers of antioxidant activity, including TAC and SOD. The values in the following Outcome Measure Data Table refer to the means of measurements at 4 follow-ups.
Time Frame: Blood samples are obtained at the end of each round of 4 follow-ups with an interval of 2 weeks in the last 2 months of intervention.
Measure: Mean (Standard Deviation); unit: U/ml
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
Number analyzed (Participants) | 34 | 31
U/ml
  TAC | 6.09 (2.15) | 5.80 (2.36)
  SOD | 364.34 (42.69) | 356.59 (43.90)

2. Primary Outcome: Biomarkers of Inflammation-Interleukin-6 (IL-6) and Tumour Necrosis Factor-α (TNF-α)
Description: 2 inflammatory biomarkers in our study including IL-6 and TNF-α are measured. The values in the following Outcome Measure Data Table refer to the means of measurements at 4 follow-ups.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
Number analyzed (Participants) | 34 | 31
pg/ml
  IL-6 | 0.72 (0.63) | 1.76 (5.75)
  TNF-α | 0.35 (0.47) | 0.54 (1.42)

3. Primary Outcome: Cogulation Biomarker-von Willebrand Factor (vWF)
Description: We measure vWF level in serum, one of the measured cogulation biomarkers in our study. The values in the following Outcome Measure Data Table refer to the means of measurements at 4 follow-ups.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mIU/ml
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
Number analyzed (Participants) | 34 | 31
mIU/ml | 1669.70 (1022.98) | 2144.30 (1674.32)

4. Primary Outcome: Biomarkers of Endothelial Function and Stress Hormone
Description: We measure endothelial function biomarkers, including E-selectin and endothelial nitric oxide synthase (eNOS), and 4 stress hormones, including corticotropin releasing hormone (CRH), adrenocorticotropic hormone (ACTH), cortisol and serotonin. The values in the following Outcome Measure Data Table refer to the means of measurements at 4 follow-ups.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
Number analyzed (Participants) | 34 | 31
ng/ml
  E-selectin | 12.23 (5.38) | 14.16 (6.81)
  eNOS | 5.99 (9.19) | 4.29 (7.55)
  CRH | 2.96 (0.48) | 3.06 (0.47)
  Cortisol | 168.01 (48.62) | 184.49 (68.42)
  ACTH | 0.34 (0.10) | 0.39 (0.12)
  serotonin | 153.56 (63.89) | 151.17 (61.63)

5. Primary Outcome: Endothelial Function Biomarker-Endothelin-1(ET-1)
Description: We measure ET-1 level in serum, an endothelial function biomarker. The values in the following Outcome Measure Data Table refer to the means of measurements at 4 follow-ups.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
Number analyzed (Participants) | 34 | 31
pg/ml | 1.80 (2.26) | 2.82 (4.92)

6. Primary Outcome: Cogulation Biomarker-Fibrinogen
Description: We measure the serum level of fibrinogen, one of the two measured cogulation biomarkers in our study. The values in the following Outcome Measure Data Table refer to the means of measurements at 4 follow-ups.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg/ml
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
Number analyzed (Participants) | 34 | 31
µg/ml | 2.25 (1.06) | 2.63 (1.28)

7. Primary Outcome: High-sensitivity C-reactive Protein (Hs-CRP)-an Inflammatory Biomarker
Description: The serum levels of hs-CRP are measured. The values in the following Outcome Measure Data Table refer to the means of measurements at 4 follow-ups.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg/ml
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
Number analyzed (Participants) | 34 | 31
µg/ml | 12.81 (19.91) | 19.93 (30.03)

8. Primary Outcome: Oxidized Low Density Lipoprotein (Ox-LDL)-an Oxidative Stress Biomarker
Description: Peripheral blood samples (5 ml) were drawn, separated into serum, and stored at -80 ℃ within 30 minutes. We measure the serum level of ox-LDL. The values in the following Outcome Measure Data Table refer to the means of measurements at 4 follow-ups.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
Number analyzed (Participants) | 34 | 31
U/L | 34.74 (9.85) | 40.11 (22.83)

9. Primary Outcome: Glutathione Peroxidase (GSH-Px)-a Biomarker of Antioxidant Activity
Description: Peripheral blood samples (5 ml) were drawn, separated into serum, and stored at -80 ℃ within 30 minutes. We also measure GSH-Px. The values in the following Outcome Measure Data Table refer to the means of measurements at 4 follow-ups.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mU/ml
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
Number analyzed (Participants) | 34 | 31
mU/ml | 625.95 (157.42) | 581.51 (171.92)

10. Primary Outcome: Serum Level of Lipid Peroxidation (LPO)-a Biomarker of Oxdative Stress
Description: Peripheral blood samples (5 ml) were drawn, separated into serum, and stored at -80 ℃ within 30 minutes. We measure the serum level of LPO. The values in the following Outcome Measure Data Table refer to the means of measurements at 4 follow-ups.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg/ml
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
Number analyzed (Participants) | 34 | 31
µg/ml | 0.54 (0.15) | 0.58 (0.17)

11. Secondary Outcome: Blood Pressure
Description: After sitting in a quiet room for at least 5 min, participants had their left upper arm blood pressure measured by trained technicians using an electronic sphygmomanometer at least three times with 3-min minimum intervals between measurements. The second and third sets of readings were averaged to obtain systolic BP (SBP) and diastolic BP (DBP). If the differences among the three measurements were bigger than 5 mmHg, a new round of measurements was arranged. The values in the following Outcome Measure Data Table refer to the means of measurements at 4 follow-ups.
Time Frame: Blood pressure are measured at the end of each round of 4 follow-ups with an interval of 2 weeks in the last 2 months of intervention.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
Number analyzed (Participants) | 34 | 31
mmHg
  SBP | 110.01 (11.39) | 111.55 (10.89)
  DBP | 67.20 (6.05) | 67.29 (7.97)

12. Secondary Outcome: Insulin Resistance
Description: The biomarker of insulin resistance is measured, calculated by fasting glucose and fasting insulin using the formula of [fasting insulin (mU/L) × fasting glucose (mmol/L)]/22.5. The values in the following Outcome Measure Data Table refer to the means of measurements at 4 follow-ups.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L × mU/L
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
Number analyzed (Participants) | 34 | 31
mmol/L × mU/L | 1.40 (0.94) | 1.42 (0.91)

13. Secondary Outcome: Skin Inflammation Biomarkers
Description: 2 infammation biomarkers from skin samplings are measured, including interleukin-1 Alpha (IL-1α) and Interleukin-1 receptor antagonist (IL-1Rα). The values in the following Outcome Measure Data Table refer to the means of measurements at 4 follow-ups.
Time Frame: Skin samplings are obtained at the end of each round of 4 follow-ups with an interval of 2 weeks in the last 2 months of intervention.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
Number analyzed (Participants) | 34 | 31
pg/ml
  IL-1α | 184.49 (107.31) | 230.90 (163.97)
  IL-1Rα | 54.00 (93.48) | 42.00 (119.54)

14. Secondary Outcome: Skin Oxidative Stress Biomarker-Carbonyl Protein
Description: oxidative stress biomarker in skin samplings includes carbonyl protein. The values in the following Outcome Measure Data Table refer to the means of measurements at 4 follow-ups.
Time Frame: Skin samplings are obtained at the end of each round of 4 follow-ups with an interval of 2 weeks in the last 2 months.
Measure: Mean (Standard Deviation); unit: µg/ml
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
Number analyzed (Participants) | 34 | 31
µg/ml | 35.93 (15.37) | 44.89 (24.01)

15. Secondary Outcome: Lung Function-Forced Vital Capacity (FVC) and Forced Expiratory Volume in 1 Second (FEV1)
Description: Indicators of lung function include forced vital capacity (FVC) and andforced expiratory volume in 1 second (FEV1). The values in the Outcome Measure Data Table refer to the means of measurements at 4 follow-ups.
Time Frame: Lung function is measured at the end of each round of 4 follow-ups with an interval of 2 weeks in the last 2 months of intervention.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
Number analyzed (Participants) | 34 | 31
L
  FVC | 3.18 (0.48) | 3.16 (0.62)
  FEV1 | 3.75 (0.64) | 3.73 (0.87)

16. Secondary Outcome: Lung Function-Peak Expiratory Flow (PEF)
Description: Additional indicator of lung function includes peak expiratory flow (PEF). The values in the Outcome Measure Data Table refer to the means of measurements at 4 follow-ups.
Time Frame: as for outcome 15
Measure: Mean (Standard Deviation); unit: L/s
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
Number analyzed (Participants) | 34 | 31
L/s | 6.55 (1.44) | 6.38 (1.60)

17. Secondary Outcome: Skin Antioxidant Biomarker-Total Antioxidant Capacity (TAC)
Description: we measure TAC level, an antioxidant biomarker in skin samplings. The values in the following Outcome Measure Data Table refer to the means of measurements at 4 follow-ups.
Time Frame: Skin samplings are obtained at the end of each round of 4 follow-ups with an interval of 2 weeks in the last 2 months.
Measure: Mean (Standard Deviation); unit: nmol/mL
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
Number analyzed (Participants) | 34 | 31
nmol/mL | 42.99 (95.34) | 35.73 (17.55)

18. Secondary Outcome: Skin Antioxidant Biomarker-Glutataione (GSH)
Description: we measure another skin antioxidant biomarker-GSH, . The values in the following Outcome Measure Data Table refer to the means of measurements at 4 follow-ups.
Time Frame: Skin samplings are obtained at the end of each round of 4 follow-ups with an interval of 2 weeks in the last 2 months.
Measure: Mean (Standard Deviation); unit: ppb
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
Number analyzed (Participants) | 34 | 31
ppb | 2.21 (1.70) | 0.42 (1.07)

19. Post Hoc Outcome: Differences in Metabolite Levels Detected in Serum Metabolomics Between the Two Groups
Description: Mass spectrometry-based serum metabolomics is non-targeted. The study is to find the differential metabolites in serum between fish oil and placebo groups.
Time Frame: as for outcome 1
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: At the end of week 8, week 10, week 12 and week 14 during the period of supllementation
Arm/Group | Fish Oil Supplementation | Sunflower Seed Oil Supplementation
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/31
Other Adverse Events (participants affected / at risk) | 0/34 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT03255187/Prot_SAP_000.pdf